CLINICAL TRIAL: NCT04176562
Title: Prospective Study on Safety and Performance of Surgalign spINE Products
Brief Title: Prospective SPINE Registry
Acronym: SPINE
Status: Recruiting | Type: Observational
Sponsor: Xtant Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: 19094
Record Dates: First submitted 2019-11-20; First posted 2019-11-25 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Sacroiliac; Fusion; Sacroiliac; Joint Diseases; Musculoskeletal Diseases; Spinal Disease; Spinal Stenosis; Spinal Instability; Fusion of Joint; Fusion of Spine; Spinal Fusion; Spine
MeSH Terms: conditions — Joint Diseases; Musculoskeletal Diseases; Spinal Diseases; Spinal Stenosis; Ankylosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: RTI Spine products — * Interbody fusion devices - intended to help facilitate fusion by providing a platform for bone growth, while maintaining height and decompression.
  * Supplemental fixation and/or stabilization devices - are intended to stabilize the spine to allow for fusion to occur, maintain current spinal movement, correct deformities or curvature, treat trauma, spinal stenosis, tumor and pseudarthrosis.
  * Bone graft substitute - is intended to aid in fusion.

SUMMARY:
This study is a prospective, multi-center, open label registry designed to collect real-world data on performance and safety data on RTI's spine products.

ELIGIBILITY:
Inclusion Criteria:

1. Candidate for RTI spine product.
2. Willing and able to consent to the study.

Exclusion Criteria:

1. Patient who is, or is expected to be inaccessible for follow-up.
2. Patient meets any exclusion criteria required by local law (e.g. age, mental capacity, etc.).
3. Other concurrent medical or other condition (chronic or acute in nature) that in the opinion of the investigator may prevent participation or otherwise render patient ineligible for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that have spinal problems requiring treatment with an RTI Surgical spine product.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2020-01-28 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Intervention Rates | 1 month, 3 months, 6 months, 12 months, and 24 months
  Rates of reoperation and/or revision procedures at index level

SECONDARY OUTCOMES:
Fusion | 1 month, 3 months, 6 months, 12 months, and 24 months
  Fusion success measures by radiological assessment (x-ray, CT scan, MRI, etc.)
Radiographic Findings | 1 month, 3 months, 6 months, 12 months, and 24 months
  Change in radiographic findings
Adverse Events | 1 month, 3 months, 6 months, 12 months, and 24 months
  Number of procedure and device related adverse events
Disability (Cervical) | 1 month, 3 months, 6 months, 12 months, and 24 months
  Change in Neck Disability Index
Disability (non-Cervical) | 1 month, 3 months, 6 months, 12 months, and 24 months
  Change in Oswestry Disability Index
Pain Change | 1 month, 3 months, 6 months, 12 months, and 24 months
  Change in pain as determined by Visual Analogue Scale (VAS)
Time to Intervention | 1 month, 3 months, 6 months, 12 months, and 24 months
  Time to first reoperation and/or revision procedure at index leve

CONTACTS AND LOCATIONS:
Locations (12):
- United States (7):
  - Hartford Hospital, Hartford, Connecticut
  - Florida Back Institute, Boca Raton, Florida
  - Spine Institute of South Florida, Delray Beach, Florida
  - Suburban Orthopaedics, Bartlett, Illinois
  - Indiana Spine Group, Carmel, Indiana
  - DK Orthopedics, Crown Point, Indiana
  - Lindner Center for Research & Education at The Christ Hospit, Cincinnati, Ohio
- Germany (4):
  - STENUM Ortho Fachklinik, Ganderkesee
  - Wirbelsäulenzentrum Fulda | Main | Kinzig, Gelnhausen
  - Katholisches Klinikum Koblenz - Montabaur, Koblenz
  - St. Christopherus Krankenhaus - Katholisches Klinikum, Werne
- Hospital Nacional de Parapléjicos, Toledo, Spain

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD